CLINICAL TRIAL: NCT00988377
Title: The Effect of Whey Protein on Short-term Food Intake and Post-meal Blood Glucose Response in Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Mondelēz International, Inc. (Industry)
Responsible Party: Dr. G. Harvey Anderson, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Kraft_whey protein: study 1
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Prevention; Obesity Prevention
Keywords: whey protein; subjective appetite; shor-term food intake; blood glucose
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 10 g whey protein (Experimental)
  Interventions: Other: dietary intervention
- 20 g whey protein (Experimental)
  Interventions: Other: dietary intervention
- 30 g whey protein (Experimental)
  Interventions: Other: dietary intervention
- 40 g whey protein (Experimental)
  Interventions: Other: dietary intervention
- water control (Experimental): Iso-volumetric (300 ml) water control (Crystal Springs, Canada)
  Interventions: Other: water control

INTERVENTIONS:
Other: dietary intervention — whey protein 10-40 g
  Arms: 10 g whey protein; 20 g whey protein; 30 g whey protein; 40 g whey protein
Other: water control — Iso-volumetric (300 ml) water control (Crystal Springs, Canada)
  Arms: water control

SUMMARY:
The objective of this study was to describe relationships among whey protein when consumed before a meal on food intake and pre- and post-meal satiety, blood glucose in healthy young adults.

DETAILED DESCRIPTION:
A randomized, cross-over design study was conducted. Whey protein preloads (10-40 g) were provided in 300 ml water. At 30 min following consumption, subjects were fed an ad libitum pizza meal. Satiety, and blood glucose were measured at baseline and selected intervals pre- (0, 15 and 30 min) and post-meal (50, 65, 80 and 95 min).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normal weight ( 18-24.9 kg/m²)
* young aged 20-27 year old

Exclusion Criteria:

* breakfast skippers
* smokers
* dieters
* individuals with diabetes (fasting BG ≥ 7.0 mmol/L) or other metabolic diseases

Ages: 20 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Blood glucose subjective appetite Food intake at 30 min | 0-95 min

SECONDARY OUTCOMES:
physical comfort palatability | 0-95 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Department of Nutritional Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Akhavan T, Luhovyy BL, Brown PH, Cho CE, Anderson GH. Effect of premeal consumption of whey protein and its hydrolysate on food intake and postmeal glycemia and insulin responses in young adults. Am J Clin Nutr. 2010 Apr;91(4):966-75. doi: 10.3945/ajcn.2009.28406. Epub 2010 Feb 17. PMID 20164320